CLINICAL TRIAL: NCT05638880
Title: Clinical Study to Evaluate the Possible Efficacy and Safety of Levocetirizine in Patients With Diabetic Kidney Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mostafa Bahaa (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Mostafa Bahaa, Teaching Assistant, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS.21.21.1776
Record Dates: First submitted 2022-11-28; First posted 2022-12-06 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Valsartan; empagliflozin; levocetirizine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): 30 patients will receive Valsartan 80 mg once daily titrated till blood pressure ≤ 130/80 plus Empagliflozin 10 mg once daily for 3 months
  Interventions: Drug: Valsartan 80 mg; Drug: Empagliflozin 10 MG
- Levocetirizine group (Active Comparator): 30 patients will receive Valsartan 80 mg once daily titrated till blood pressure ≤ 130/80 plus Empagliflozin 10 mg once daily plus Levocetirizine 5 mg once daily in the evening titrated according to creatinine clearance for 3 months.
  Interventions: Drug: Valsartan 80 mg; Drug: Empagliflozin 10 MG; Drug: Levocetirizine

INTERVENTIONS:
Drug: Valsartan 80 mg — Valsartan is an angiotensin receptor blocker.
Drug: Empagliflozin 10 MG — Empagliflozin is an oral hypoglycemic drug.
Drug: Levocetirizine — Levocetirizine, Histamine-1 receptor antagonists provide a highly successful approach for controlling allergic and inflammatory conditions
  Arms: Levocetirizine group

SUMMARY:
The prevalence of diabetes mellitus is increasing worldwide, and its complications are one of the leading causes of mortality from non-communicable diseases. Due to the high prevalence of diabetes and because 30-40% of diabetic patients [both type 1 (T1DM) and type 2 (T2DM) diabetes mellitus] develop kidney dysfunction, diabetic nephropathy (DN) is the main cause of end-stage renal disease worldwide. The renin-angiotensin-aldosterone system (RAAS), endothelin, and urotensin II are vasoactive hormones that have been extensively studied as other mediators although their relation to diabetic nephropathy is still speculative.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 65.
* Both genders will be included.
* Type II diabetes mellitus confirmed by Glycosylated Hemoglobin A₁C.
* Diagnosis of diabetic nephropathy, which will be defined as persistent albuminuria with urinary albumin creatinine ratio (UACR) range [30-300 mg /gm], confirmed on at least two occasions 3-6 months apart, with or without decline in glomerular filtration rate at screening and receiving angiotensin receptor blockers (ARBs) and sodium-glucose cotransporter 2 (SGLT2) inhibitors therapy.
* Hemoglobin A₁C ranges from 6.5% to 10% with regular use of insulin and or/oral hypoglycemic drugs.

Exclusion Criteria:

* Other types of diabetes mellitus
* Uncontrolled hypertension (Blood pressure ≥ 180/110).
* Urinary tract infection.
* Severe anemia (Hemoglobin ˂10).
* Critically ill patient.
* Past operation, past history of trauma, heavy exercise.
* Severe renal failure (e GFR ˂ 30ml/min/1.73 m2).
* Systemic inflammatory and autoimmune diseases.
* Malignancy.
* Pregnancy and lactating women.
* Other causes of chronic kidney disease.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
Reduction of albuminuria | 3 months
  Reduction of albuminuria in diabetic nephropathy

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Derived] Rizk MA, El-Haggar SM, Ibrahim OM, Ghazi HA. Efficacy of levocetirizine in reducing albuminuria and inflammatory biomarkers in patients with diabetic kidney disease: A randomized controlled trial. J Diabetes Complications. 2025 Nov;39(11):109175. doi: 10.1016/j.jdiacomp.2025.109175. Epub 2025 Sep 10. PMID 40946347